CLINICAL TRIAL: NCT05383963
Title: Evaluation of Parameters Collected From Routine Data for the Diagnosis of Sepsis and Septic Shock and Their Influence on Time to Diagnosis and Patient Outcome (QUICK-SEPSIS)
Brief Title: Evaluation of Parameters Collected From Routine Data for the Diagnosis of Sepsis and Septic Shock and Their Influence on Time to Diagnosis and Patient Outcome
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative Intensive Care Medicine CCM/CVK, Charité - Universitätsmedizin Berlin, Charite University, Berlin, Germany
Other Study IDs: QUICK-SEPSIS
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective observational study to develop a Machine Learning Algorithm to evaluate parameters collected from routine data for the diagnosis of sepsis and septic shock and their influence on time to diagnosis and patient outcome.

DETAILED DESCRIPTION:
Retrospective routine data from the medical records of the department of anesthesiology and operative intensive care from 01. 01. 2007 to 31. 12. 2021 are analyzed in digital form.

The first step is the development of a machine learning algorithm (MLA). This MLA will be validated and analyzed for his predictive value with regard to early diagnosis of sepsis/septic shock depending on the conceptual value of detection variables (Sepsis-3 vs. SIRS). Further analysis will focus on improvement of accuracy for the MLA and the effect of these detection variables on quality of treatment processes and also on economic consequences like cost and revenue.

Timeline:

1. Conception and development of the ML Algorithm (6 months)
2. Identification and diagnostic validation of sepsis patients (6 months)
3. Secondary analyses (36 months)

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* ICU stay of > 24 hours

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care unit patients (female, male, miscellaneous) from the age of 18 years with an intensive care stay of > 24 hours in an intensive care unit since 01. 01. 2007 from the Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK)
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Sepsis/septic shock | 01.01.2007 -31.12.2021
  Development of a machine learning algorithm (MLA) for the prediction of sepsis/septic shock from hospital routine data.

SECONDARY OUTCOMES:
Predictive accuracy | 01.01.2007 -31.12.2021
  Evaluation of the predictive accuracy (= predictive value) of the respective sepsis diagnostic algorithm (i.e. comparison of the concepts SIRS and Sepsis-3)
Diagnostic accuracy | 01.01.2007 -31.12.2021
  Identification of additional variables for diagnostic accuracy (laboratory values, clinical parameters and vital-sign monitor parameters and other relevant health data
Performance indicators | 01.01.2007 -31.12.2021
  Evaluation of performance indicators of clinical routine processes (Intensive care quality indicators)
Case costs | 01.01.2007 -31.12.2021
  Case costs related to hospitalization
Revenues | 01.01.2007 -31.12.2021
  Revenues related to hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine CCM/CVK, Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No